CLINICAL TRIAL: NCT04964414
Title: Prospective Randomized Study of the Treatment of Pediatric Patients That Lost Sense of Smell Due to COVID-19
Brief Title: Treatment of Pediatric Patients That Lost Sense of Smell Due to COVID-19
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Amanda Stapleton (Other)
Responsible Party: Sponsor-Investigator, Amanda Stapleton, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY21050012
Record Dates: First submitted 2021-07-15; First posted 2021-07-16 (Actual); Results first posted 2024-02-08 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Dysosmia; Anosmia; Covid19
Keywords: Sino-Nasal Outcome Test; Smell Test
MeSH Terms: conditions — Olfaction Disorders; Anosmia; COVID-19 | interventions — Olfactory Training; Budesonide

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Smell Retraining Only (Active Comparator): Participants will undergo smell retraining for 8 weeks. Each week, participants will choose 4 scents. They will smell each item for 15 seconds very close to the nose once a day.
  Interventions: Other: Smell Retraining
- Smell Retraining + Budesonide (Experimental): Participants will undergo smell retraining as described above. They will also complete budesonide irrigations once a day by pouring 0.5mg/2ml of budesonide into a irrigation bottle with saline and irrigating the nose.
  Interventions: Other: Smell Retraining; Drug: Budesonide

INTERVENTIONS:
Other: Smell Retraining — Smell practice with household scented items
  Other Names: Smell Training; Olfactory Retraining
Drug: Budesonide — Nasal irrigation with liquid steroid
  Other Names: Nasal Glucocorticoid Irrigation
  Arms: Smell Retraining + Budesonide

SUMMARY:
This research study is a randomized controlled trial in pediatric and young adult patients who have lost their sense of smell due to COVID-19 viral infection. The goals are:

1. to learn more about the effects of smell retraining therapy on smell loss following COVID-19 and
2. to determine if budesonide-saline irrigations make smell retraining therapy more effective.

DETAILED DESCRIPTION:
Researchers will screen all potentially eligible patients that have 'loss of smell' as their reason for visit at UPMC Children's Hospital of Pittsburgh Division of Pediatric Otolaryngology.

At the initial consult appointment at the Division of Pediatric Otolaryngology, listed study team members will perform a smell identification test called the UPSIT (University of Pennsylvania Smell Identification Test) and give the SNOT-22 (Sino-Nasal Outcome Test-22) survey. The UPSIT is a 40-item scratch and sniff test with a four-choice multiple choice question on each of the 10 pages in the booklet. Indication of smell loss can be determined - anosmia (total loss) and mild, moderate, or severe microsomia and a detection for malingering. The SNOT-22 is a 22 question survey that asks about symptoms and social/emotional consequences of a nasal disorder. The survey is on a 6 point scale - No problem (0), very mild problem (1), mild or slight problem (2), moderate problem (3), severe problem (4), and problem as bad as it can be (5).

A randomized clinical trial will be performed with two arms for those that have lost their sense of smell for at least 8 weeks: 1) smell retraining for 8 weeks 2) smell retraining + Budesonide irrigations for 8 weeks. Smell retraining consists of choosing 4 scents each week and smelling each item for 15 seconds very close to the nose once a day. Budesonide irrigations will be done once a day by pouring 0.5mg/2ml of Budesonide into a irrigation bottle with saline and irrigating the nose. Participants may do the therapies at any point during the day.

Children and young adults ages 6 to 21 will be enrolled with 30 children block randomized in each arm, in which up to 10 children in each arm will be those who did not have a positive COVID-19 antigen test or confirmed COVID-19 by history. COVID-19 testing will be used for randomization purposes, but will not be limited to testing due to the inclusion of confirmation by history.

Two groups of subjects for study inclusion:

Group 1:

COVID-19 by clinical history or lab testing (n=40 (20 randomized to each group)) Those with COVID-19 confirmation by clinical history may not have had a COVID-19 positive test.

Group 2:

Those that did not have COVID-19 by clinical history or lab testing (n=20 (10 randomized to each group)) These subjects may have had a negative COVID-19 test or no clinical history of COVID-19.

Each child, with the help of their parents, will do the assigned therapy and fill out a daily Smell Diary. The child will pick 4 scents each week to perform the smell retraining each day that week. The child or parent will check mark every day that the 4 scents were smelled. The scents do not have to be new each week. Once a week the child will rate their loss of smell on a scale from 0 (no loss) to 10 (total loss).

Researchers will check in with the parent or participant on weeks 3, 5, and after the 8 week period. Families will return the Smell Diary at their standard of care follow-up appointment at 8 weeks (range 8 to 12 weeks). The UPSIT and the SNOT-22 will be given at the follow-up appointment. If the participants' sense of smell did not return to baseline at the follow-up, they will be asked to return at 6 months after the initial consult. If the participants' sense of smell has still not returned at the 6 month appointment, they will be asked to follow-up at 1 year after the initial consult. The UPSIT and SNOT-22 will be given at each of these appointments. If smell was not a baseline at 8 weeks, listed investigators will call the subject or subjects' parents at 6 months and 1 year after the initial appointment to check-in and for a reminder to schedule a follow-up appointment.

If participants do not have an 8-week follow-up visit, they may be mailed an UPSIT to complete at home and return by mail. They may also complete the SNOT-22 by mail or phone, and they may return the smell diary by email.

If patients were initially randomized to the smell retraining only, after the initial 8-12 weeks of therapy they may be prescribed budesonide as part of standard of care to maximize medical management as needed. We will invite participants to fill out a new smell diary during this time and we will collect any data available from the smell diary, UPSIT, and SNOT-22 at their standard of care visit after 8-12 weeks of budesonide irrigation. Patients who have already completed more than 12 weeks of smell retraining will not be included in this arm; although budesonide may be prescribed based on physician discretion, data will not be collected following budesonide treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ages 6 to 21 who have loss of smell (anosmia) or dysosmia (disordered smell perception) and thought to have occurred due to COVID-19.
* Subjects who are able to complete the smell test (UPSIT), self-report their loss of smell, and do the assigned daily therapy.

Exclusion Criteria:

* Duration of anosmia or dysosmia <60 days
* Previous smell retraining
* Prior interventions for loss of smell (excluding those on Flonase and Azelastine)
* Contraindications for nasal budesonide treatment, as determined by the treating physician
* Active cigarette smoker or use of vapes
* Previous head trauma
* Congenital anosmia
* History of brain tumor
* Neurocognitive disorders
* Multiple sclerosis
* Seizure disorder
* Cystic fibrosis
* Primary Ciliary Dyskinesia
* History of nasal polyps
* Inability to self-report

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda L Stapleton, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) may be shared, after de-identification, with researchers who provide a methodologically sound proposal. IPD to be shared will include that necessary to achieve the aims in the approved proposal.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 1 year after publication of summary data. Ending 5 years after publication.
Access Criteria: Proposals should be directed to shafferad@upmc.edu. To gain access, data requestors will need to sign data access agreement.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant was placed in a treatment arm (OT + BI) different than what was randomly assigned (OT) at the initial clinic visit.
Period: Overall Study
Arm/Group | Smell Retraining Only | Smell Retraining + Budesonide
Started | 11 | 9
8-12 Week Follow-up | 7 | 1
6 Month Follow-up (Budesonide was added to smell retraining for one of these patients at time of the 8-12 week follow-up visit.) | 3 | 0
12 Month Follow-up | 0 | 0
Completed | 0 | 0
Not Completed | 11 | 9
Not completed — Lost to Follow-up | 10 | 8
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Smell Retraining Only | Smell Retraining + Budesonide | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Continuous [Median (Full Range); unit: years] | 13 [7 to 19] | 16 [14 to 17] | 16 [7 to 19]
Age, Customized [Count of Participants; unit: Participants]
  7-12 years | 5 | 0 | 5
  13-18 years | 6 | 9 | 15
  19-21 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 8 | 19
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 10 | 8 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Primary Complaint [Count of Participants; unit: Participants] — Primary compliant at initial clinic visit
  Participants
    Abnormal Smell and Taste | 6 | 8 | 14
    Abnormal Smell Only | 5 | 1 | 6
Symptom Onset Post-COVID-19 [Count of Participants; unit: Participants]
  Immediate | 7 | 7 | 14
  Delayed | 2 | 2 | 4
  Unknown | 2 | 0 | 2
Medical History [Count of Participants; unit: Participants]
  Allergic Rhinitis: Yes | 0 | 3 | 3
  Allergic Rhinitis: No | 11 | 6 | 17
  Environmental Allergies: Yes | 0 | 3 | 3
  Environmental Allergies: No | 11 | 6 | 17
  Immunosuppression: Yes | 1 | 1 | 2
  Immunosuppression: No | 10 | 8 | 18
  Deviated Septum: Yes | 0 | 1 | 1
  Deviated Septum: No | 11 | 8 | 19
  History of Radiation: Yes | 0 | 1 | 1
  History of Radiation: No | 11 | 8 | 19
Vaccinated against COVID-19 [Count of Participants; unit: Participants]
  Yes | 2 | 0 | 2
  No | 2 | 1 | 3
  Unknown | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in University of Pennsylvania Smell Identification Test (UPSIT) Score From Baseline to First Follow-up
Description: Change in University of Pennsylvania Smell Identification Test (UPSIT) score from baseline at the initial consult appointment to the first follow-up appointment at 8 weeks (range 8 to 12 weeks). The UPSIT is a smell identification test and is a 40-item scratch and sniff test with a four-choice multiple choice question on each of the 10 pages in the booklet. Indication of smell loss can be determined - anosmia (total loss) and mild, moderate, or severe microsomia and a detection for malingering. The minimum possible score is a 0 and the maximum is a 40. A higher score indicates better smell/outcome.
Time Frame: Before and after 8-12 weeks of smell retraining
Population: Patients who completed 8-12 week follow-up assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Smell Retraining Only | Smell Retraining + Budesonide
Number analyzed (Participants) | 7 | 1
score on a scale
  Before smell retraining | 23.3 (7.3) | 34
  After 8-12 weeks of smell retraining | 22.3 (7.3) | 35
Statistical Analysis 1: Comparison: Smell Retraining Only; Test type: Superiority; p = 0.6, Paired t-test

2. Secondary Outcome: Change in Sino-nasal Outcome Test-22 (SNOT-22) Score From Baseline to First Follow-up
Description: Change in Sino-nasal Outcome Test-22 (SNOT-22) score from baseline at the initial consult appointment to the first follow-up appointment at 8 weeks (range 8 to 12 weeks). The SNOT-22 is a 22 question survey that asks about symptoms and social/emotional consequences of a nasal disorder. The survey is on a 6 point scale - No problem (0), very mild problem (1), mild or slight problem (2), moderate problem (3), severe problem (4), and problem as bad as it can be (5). The minimum possible score is 0 and the maximum is 110. A higher score indicates more sino-nasal symptoms/worse outcome.
Time Frame: Before and after 8-12 weeks of smell retraining
Population: Patients who completed 8-12 week follow-up assessments
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Smell Retraining Only | Smell Retraining + Budesonide
Number analyzed (Participants) | 7 | 1
score on a scale
  Before smell retraining | 23 [10 to 41] | 37
  After 8-12 weeks of smell retraining | 25 [11 to 37] | 39
Statistical Analysis 1: Comparison: Smell Retraining Only; Test type: Superiority; p = 0.6, Wilcoxon signed-rank

3. Secondary Outcome: Change in Loss of Smell Question Score From Baseline to First Follow-up
Description: Change in loss of smell on a 0-10 scale from baseline at the initial consult appointment to the first follow-up appointment at 8 weeks (range 8 to 12 weeks). Subjects are asked to rate the symptom severity of loss of smell from 0 (no loss) to 10 (total loss). A higher score indicates worse smell/outcome.
Time Frame: Before and after 8-12 weeks of smell retraining
Population: Patients who returned the smell diary and completed the loss of smell scale before and after 8-12 weeks of smell retraining
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Smell Retraining Only | Smell Retraining + Budesonide
Number analyzed (Participants) | 5 | 1
score on scale
  Before smell retraining | 6.0 (3.3) | 6.0
  After 8-12 weeks of smell retraining | 5.0 (3.7) | 8.0
Statistical Analysis 1: Comparison: Smell Retraining Only; Test type: Superiority; p = 0.09, Paired t-test

4. Secondary Outcome: Change in University of Pennsylvania Smell Identification Test (UPSIT) Score From Baseline to 6 Month Follow-up
Description: Change in University of Pennsylvania Smell Identification Test (UPSIT) score from baseline at the initial consult appointment to the 6 month follow-up appointment. The minimum possible score is a 0 and the maximum is a 40. A higher score indicates better smell/outcome.
Time Frame: Baseline and 6 months after initial consult appointment
Population: Patients who completed 6 month follow-up assessments
Measure: Median (Full Range); unit: score on scale
Arm/Group | Smell Retraining Only | Smell Retraining + Budesonide
Number analyzed (Participants) | 3 | 0
score on scale
  Before smell retraining | 15 [13 to 21] |
  After 6 months of smell retraining | 17 [14 to 24] |

5. Secondary Outcome: Change in Sino-nasal Outcome Test-22 (SNOT-22) Score From Baseline to 6 Month Follow-up
Description: Change in Sino-nasal Outcome Test-22 (SNOT-22) score from baseline at the initial consult appointment to the 6 month follow-up appointment. The minimum possible score is 0 and the maximum is 110. A higher score indicates more sino-nasal symptoms/worse outcome.
Time Frame: Baseline and 6 months after initial consult appointment
Population: Patients who completed 6 month follow-up assessments
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Smell Retraining Only | Smell Retraining + Budesonide
Number analyzed (Participants) | 3 | 0
score on a scale
  Before smell retraining | 25 [15 to 41] |
  After 6 months of smell retraining | 9 [8 to 14] |

6. Secondary Outcome: Change in University of Pennsylvania Smell Identification Test (UPSIT) Score From Baseline to 12 Month Follow-up
Description: Change in University of Pennsylvania Smell Identification Test (UPSIT) score from baseline at the initial consult appointment to the 12 month follow-up appointment. The minimum possible score is a 0 and the maximum is a 40. A higher score indicates better smell/outcome.
Time Frame: Baseline and 12 months after initial consult appointment
Population: Patients who completed 12 month follow-up assessments
Arm/Group | Smell Retraining Only | Smell Retraining + Budesonide
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in Sino-nasal Outcome Test-22 (SNOT-22) Score From Baseline to 12 Month Follow-up
Description: Change in Sino-nasal Outcome Test-22 (SNOT-22) score from baseline at the initial consult appointment to the 12 month follow-up appointment. The minimum possible score is 0 and the maximum is 110. A higher score indicates more sino-nasal symptoms/worse outcome.
Time Frame: Baseline and 12 months after initial consult appointment
Population: Patients who completed 12 month follow-up assessments
Arm/Group | Smell Retraining Only | Smell Retraining + Budesonide
Number analyzed (Participants) | 0 | 0

8. Other Pre Specified Outcome: Change in Loss of Taste Question Score From Baseline to First Follow-up
Description: Change in loss of taste on a 0-10 scale from baseline at the initial consult appointment to the first follow-up appointment at 8 weeks (range 8 to 12 weeks). Subjects are asked to rate the symptom severity of loss of taste from 0 (no loss) to 10 (total loss). A higher score indicates less taste/worse outcome.
Time Frame: Before and after 8-12 weeks of smell retraining
Population: Patients who returned the smell diary and completed the loss of taste scale before and after 8-12 weeks of smell retraining
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Smell Retraining Only | Smell Retraining + Budesonide
Number analyzed (Participants) | 5 | 1
score on scale
  Before smell retraining | 3.6 (3.8) | 6.0
  After 8-12 weeks of smell retraining | 1.6 (2.1) | 8.0
Statistical Analysis 1: Comparison: Smell Retraining Only; Test type: Superiority; p = 0.2, Paired t-test

9. Other Pre Specified Outcome: Change in Anxiety Question Score From Baseline to First Follow-up
Description: Change in anxiety on a 0-10 scale from baseline at the initial consult appointment to the first follow-up appointment at 8 weeks (range 8 to 12 weeks). Subjects are asked to rate the symptom severity of anxiety from 0 (no anxiety) to 10 (worst possible anxiety). A higher score indicates more anxiety/worse outcome.
Time Frame: Before and after 8-12 weeks of smell retraining
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Smell Retraining Only | Smell Retraining + Budesonide
Number analyzed (Participants) | 5 | 1
score on a scale
  Before smell retraining | 5.0 (4.4) | 7.0
  After 8-12 weeks of smell retraining | 3.4 (4.4) | 8.5
Statistical Analysis 1: Comparison: Smell Retraining Only; Test type: Superiority; p = 0.2, Paired t-test

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Smell Retraining Only | Smell Retraining + Budesonide
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/9
Other Adverse Events (participants affected / at risk) | 0/11 | 0/9

LIMITATIONS AND CAVEATS:
Early termination and significant loss to follow-up leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-25): https://cdn.clinicaltrials.gov/large-docs/14/NCT04964414/Prot_SAP_000.pdf